CLINICAL TRIAL: NCT06800040
Title: Evaluating the Feasibility and Effectiveness of a Group-Based Memory Rehabilitation Program for Acquired Brain Injury (ABI) Patients
Brief Title: Testing a Group Memory Training Program for People With Brain Injuries
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Martin Kragnes Bystad, Head of research, University Hospital of North Norway
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC North ID nr. 793668; 38355/HNI0056-24 (Other: Innovation Centre, Northern Norway Regional Health Authority)
Record Dates: First submitted 2024-12-13; First posted 2025-01-29 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-01

CONDITIONS: Acquired Brain Injury (Including Stroke)
Keywords: Memory rehabilitation; Cognitive rehabilitation; Acquired brain injury; Rehabilitation after brain injury
MeSH Terms: conditions — Brain Injuries | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Memory training (Experimental)
  Interventions: Behavioral: Memory training

INTERVENTIONS:
Behavioral: Memory training — Memory training

SUMMARY:
The purpose of this study is to assess the feasibility, acceptability, and effectiveness of a 6-week group-based memory training program for individuals experiencing memory problems after acquired brain injury (ABI).

Memory impairment is a prevalent consequence of neurological disorders like stroke, traumatic brain injury (TBI), anoxia, brain tumours, or brain infections, collectively termed acquired brain injury (ABI). While memory rehabilitation has shown promise in improving cognitive function in ABI patients, individualised treatments can be resource-intensive and not readily accessible to all in need.

The program "Group-Based Memory Rehabilitation to Improve Memory for Everyday Tasks" offers an evidence-based, group-based intervention. Previous studies have demonstrated its efficacy in enhancing everyday memory function, including increased use of memory strategies, achievement of memory-related goals, and improvements in learning ability, both in the subacute and chronic phase post-injury. Furthermore, recent investigations have shown comparable efficacy when delivering the program through telehealth platforms (video conferencing).

The investigators have meticulously translated and adapted the memory program to suit Norwegian conditions. As far as the investigators are aware, this is the first time the program has undergone translation and adaptation for Norwegian speakers.

This study aims to evaluate the memory program's feasibility, acceptability, and effectiveness in a Norwegian context, aiming to support its implementation in local health services. Both physical face-to-face groups as well as telehealth delivery through videoconferencing will be evaluated. Telehealth delivery will be utilised to overcome geographical barriers and enhance accessibility for patients residing in rural or remote areas in Northern Norway, where rehabilitation services are recognized as an unmet need. A total of five groups will be run during 2025 and 2026. Three of the three groups will be digital via videoconferencing.

DETAILED DESCRIPTION:
This manualized, group-based memory intervention involves six weekly, two-hour sessions (including a break). Group sizes should be from 3 to 10 participants, as recommended by the developers, with two group leaders (psychologists/neuropsychologists). Each session encompasses education about memory and factors influencing optimal memory function, and training in the use of compensatory memory strategies (both internal strategies and external memory aids). Group exercises and discussions, as well as homework tasks between sessions, are used to facilitate learning and generalisation of memory skills. The two-hour sessions are divided into approximately 15 minutes for reviewing homework and repetition from previous sessions; 20-30 minutes for the educational component; 60-80 minutes for practising strategies and discussing their application; 10 minutes for a break. Full details of the memory intervention, including instructional guidelines, description of exercises, handouts and supporting materials, can be found in the published manual.

The memory training program will constitute a new treatment intervention in the health region of Northern Norway, and the need to carry out feasibility studies as part of the development of complex interventions has been pointed out. Hence, the objective of this study is to identify and evaluate obstacles to delivery and implementation of the program through a feasibility and acceptability study. Effectiveness of the intervention will depend on sufficient feasibility, and will also be evaluated.

The study has two aims. First, the investigators aim to explore the feasibility of delivering the intervention, and the patients acceptability of the intervention, in order to achieve optimal efficacy.

Second, the investigators will explore the effectiveness of the memory training program on participants' memory functioning.

Research question 1 What is the feasibility of the intervention, considering a) the demand for the treatment as assessed through a) Recruitment, b) Adherence, c) Acceptability by participants, and d) Format of delivery.

Research question 2 Does a group-based 6 week memory training program improve objective and subjective memory functioning in individuals with memory complaints after ABI? The aim of the program is to enhance memory functioning on one or more measures of subjective and objective memory, number of memory strategies used in daily life, and/or personal goal attainment.

ELIGIBILITY:
Inclusion Criteria:

* history of ABI (stroke/cerebrovascular incidents, traumatic brain injury, anoxia, non-progressive brain tumour, brain infection, or other non-progressive ABI) at least 6 months prior to inclusion.
* memory problems.
* sufficient Norwegian language skills to participate in assessments and group treatment.
* age between 18 and 75 years.

Exclusion Criteria:

* diagnosis of comorbid progressive neurodegenerative disorder, or serious major somatic or psychiatric conditions (e.g bipolar disorder, psychosis, severe depression)
* major cognitive impairment preventing assessment and group participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of memory training intervention: Demand for the treatment | From enrollment to the end of follow up 3 months after the intervention
  The demand for the treatment will be assessed by number of participants enrolled.
Feasibility of memory training intervention: Adherence | From enrollment to the end of follow up 3 months after the intervention
  Adherence to treatment will be measured by dropout rate.
Feasibility of memory training intervention: Acceptability by participants | From enrollment to the end of follow up 3 months after the intervention
  Acceptability by participants will be assessed through perceptions of usefulness, measured by responses to evaluation forms.
Feasibility of memory training intervention: Format of delivery | From enrollment to the end of follow up 3 months after the intervention
  Acceptability of format of delivery (face-to-face and/or telehealth attendance) will be assessed through responses to evaluation forms.

SECONDARY OUTCOMES:
Memory training effectiveness | From enrollment to the end of follow up 3 months after the intervention
  Subjective memory problems in everyday life will be measured by responses to The Everyday Memory Questionnaire - revised (EMQ-R). The EMQ-R is a 13-item scale developed as a measure of self-reported memory failures of everyday life. It is evaluated with a five-point Likert scale whereby higher scores indicate greater frequency of memory lapses.
Memory training effectiveness | From enrollment to the end of follow up 3 months after the intervention
  Subjective memory problems in everyday life will be measured by responses to the Prospective and Retrospective Memory Questionnaire (PRMQ). The Prospective and Retrospective Memory Questionnaire (PRMQ) is a self-report measure of prospective and retrospective memory slips in everyday life, which allows participants to rate the frequency of the two forms of memory failures on a five-point Likert-scale, ranging from "very often" (5) to "never" (1). It is a 16-item scale, 8 items asking about prospective memory failures, and 8 concerning retrospective memory failures.
Strategy use | From enrollment to the end of follow up 3 months after the intervention
  Description of type and number of internal and external memory strategies participants employ in their everyday life before and after the intervention, will be registered with pre- and post-evaluation forms from the published manual.
Objective verbal memory functioning | From enrollment to the end of follow up 3 months after the intervention
  Memory impairment/objective memory functioning will be assessed with standardised a neuropsychological test of verbal memory (Rey Auditory Verbal Learning Test - RAVLT).
Objective visual memory functioning | From enrollment to the end of follow up 3 months after the intervention
  Memory impairment/objective memory functioning will be assessed with a standardised neuropsychological tests of visual memory (Brief Visuospatial Memory Test-Revised - BVMT-R).
Personal memory goal | From enrollment to the end of follow up 3 months after the intervention
  Two personal memory goals will be set at baseline and self-reported attainment assessed before and after treatment using Goal Attainment Scaling (GAS). Goal attainment is rated on a 5-point scale from -2 (current level) to +2 (much more than expected). The expected level of goal attainment is scored as 0 by the participant.

OTHER OUTCOMES:
Objective attention functioning | From enrollment to the end of follow up 3 months after the intervention
  Objective attention functioning will be assessed with the Trail Making Test (TMT) A & B.
Emotional symptoms/distress | From enrollment to the end of follow up 3 months after the intervention
  Emotional distress will be measured with the Hopkins Symptoms Checklist-10 (SCL-10). The SCL-10 questionnaire employs a four-point Likert scale for each of 10 items, ranging from 1 ("not at all") to 4 ("extremely"). The scoring system is designed so that higher scores indicate increased mental health distress symptoms.
Emotional Well-being | From enrollment to the end of follow up 3 months after the intervention
  The World Health Organisation Five Well-Being Index (WHO-5) will be used to measure general well-being. The WHO-5 asks respondents to rate their interest, engagement, and mood on five questions, and the final score ranges from 0 (very poor well-being) to 100 (excellent well-being).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: Undecided